CLINICAL TRIAL: NCT04109521
Title: Milk Safety and Child Nutrition Impacts of a Training, Certification and Marketing Scheme for Informal Dairy Vendors: the MoreMilk Project, a Randomized Control Trial in Peri-urban Nairobi, Kenya
Brief Title: MoreMilk Project: Milk Safety and Child Nutrition Impacts of a Training Scheme for Dairy Vendors in Nairobi, Kenya
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The onset of the COVID-19 pandemic impeded the progression of the RCT activities as planned. Protocol activities were stopped soon after the first component of the intervention was completed.
Sponsor: The International Livestock Research Institute (ILRI) (Other)
Collaborators: International Food Policy Research Institute (Other); Bill and Melinda Gates Foundation (Other); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPP1156625
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2019-09

CONDITIONS: Food Safety; Child Nutrition
Keywords: milk safety; child; nutrition; informal sector; dairy
MeSH Terms: interventions — Certification; Marketing

STUDY DESIGN:
Intervention Model Description: A two-arm cluster-randomized, non-masked, community-based trial will be used to estimate the effectiveness of the MoreMilk intervention. A baseline and an endline survey will be done for each arm with 12 months in between; the same vendors and households will be surveyed at baseline and endline.
  The unit of randomization is a cluster of 1 to 5 vendors and the households consuming milk from those vendors. Study clusters will be randomly assigned to one of two arms: (1) Treatment arm: Training, certification, and marketing scheme for milk vendors; (2) Control arm: Delayed intervention (implemented after endline survey).
Masking Description: Due to the nature of the intervention, it will not be possible to mask allocation to the researchers and the participants. Masking will only be done at analysis stage, meaning that analysis will be done without revealing group allocation (A/B) and by someone who is not knowledgeable about the allocation of clusters to treatment or control. Masking will only be broken after the primary analyses have been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained vendors (Experimental): The intervention consists of a Training, Certification and Marketing scheme for dairy vendors operating in the informal sector. This scheme includes a 12hr training offered at the beginning of the study, followed by 2 quarterly visits where milk will be tested for microbiological quality and results will be discussed with participants.
  The training will include three main components: (i) milk hygiene and quality; (ii) business skills; (iii) milk marketing.
  Trainings will be offered free of charge. The trainings will be given by business development service (BDS) providers, who will be trained through a "training of trainers" ahead of the intervention. Quarterly visits will involve the collection of a milk sample from each participant in the experimental arm in an unannounced visit and results on the microbiological quality of the milk reported back individually and explained to each vendor.
  Interventions: Other: Training, certification and marketing
- Untrained vendors (No Intervention): Participants in the no-intervention arm will receive the same unannounced quarterly visits, where milk will be sampled and tested for microbiological quality, but results will not be shared with the participants. The participants in this arm will only receive the training upon completion of the endline survey (i.e. when the study is finished).

INTERVENTIONS:
Other: Training, certification and marketing — The 12hr training will address the vendors (i) knowledge on hygienic handling of milk, preservation and low-cost methods for testing milk safety; (ii) business skills in record keeping, access and management of credit; (iii) milk marketing. On completion of the training and successfully passing an evaluation, vendors will be given a written certificate using a format suitable to be displayed in their premises (i.e. A4 poster, a hat or badge) indicating they have completed the training. The certification will not have legal value. Two quarterly unannounced visits will be conducted to collect a milk sample from the vendors and report back the results of microbiological quality. Vendors will have access to various milk marketing and communication items to be used in their daily operations. The materials will promote milk consumption through marketing focused on messages to consumers related to (i) good milk hygiene practices, (ii) good child nutrition practices, and (iii) household diets
  Arms: Trained vendors

SUMMARY:
The objective of the MoreMilk trial is to assess the effect of a Training, Certification and Marketing intervention for milk vendors in the informal sector on the safety of the milk sold in the markets and on the nutrition of children in peri-urban areas of Kenya. The intervention is a training scheme for dairy vendors designed to improve the vendors' business skills and increase their capacity to handle milk hygienically and recognize good quality milk. It will also support vendors to adopt marketing strategies and pass on messages to their customers on the role of milk for nutrition and good food handling practices. The intervention consists of a 12hr face-to-face training, followed by quarterly visits where milk safety is tested and results are discussed with the participants. To assess the effect of this intervention on milk safety, and selected health and nutrition outcomes, the study will work with two groups of participants: dairy retailers, referred to as dairy vendors, operating in the informal sector and consumer households that purchase milk from recruited vendors. Dairy vendors will be randomly allocated to receiving the training at the beginning of the study (treatment group) or at the end of the study (control group). A baseline survey will be administered to participating vendors and households, and an endline survey will be conducted 12 months after the intervention in the same vendors and households. The vendor baseline and endline surveys will include questionnaire modules on operations, milk handling practices, and business performance. In addition, it will include a women's empowerment module to be administered to all vendors and their spouses (pro-WEAI tool). A sample of milk will also be collected to test the microbiological quality and composition of the milk. Vendors will be visited 2 additional times during the 12 months between intervention and endline, to monitor practices and business performance and to collect a milk sample to be tested for microbiological quality and milk composition. The baseline and endline surveys in households will assess milk and food expenditure, milk handling and consumption practices, and a 24hr dietary recall for the index child, as well as length/height and weight of the index child and his/her mother .

DETAILED DESCRIPTION:
The International Livestock Research Institute (ILRI), together with partners, has pioneered an approach to improving the safety of food sold in informal markets by professionalizing informal traders who operate in these markets in low- and middle-income countries. The approach involves training vendors in hygiene and business skills and improving their ability to market products through brand creation, building skills in sales and milk promotion, and/or social marketing. The approach appears sustainable and scalable, but the nutrition and health impacts, though potentially important, have not been evaluated. The objective of the study is to assess the impact of a Training, Certification and Marketing intervention for milk vendors in the informal sector on milk safety and nutrition outcomes in children in peri-urban areas of Kenya.

The study will be conducted in 3 sub-counties in peri-urban Nairobi, Kenya. The study area was selected for its peri-urban status, ongoing urbanization, and high density of livestock and dairy production. The target wards are characterized by neighborhoods with adequate infrastructure and multi-storey buildings and areas with tin-roofed houses and limited access to piped water, sanitation and electricity. Importantly, it is estimated that about 70% (Kenya Market Trust, 2016) of the milk consumed in the study area is sold through the informal dairy vendors-vendors that sell unpackaged or not-formally processed milk-who are the focus of this study.

A two-arm cluster-randomized, non-masked, community-based trial will be used to estimate the effectiveness of the MoreMilk intervention. The RCT aims at answering the following two research questions:

* Does a "training, certification and marketing" intervention for dairy vendors operating in the informal dairy markets in peri-urban Nairobi improves the microbiological quality (i.e. safety) of the unpacked milk sold in informal markets?
* Does a "training, certification and marketing" intervention for dairy vendors operating in the informal dairy markets in peri-urban Nairobi increase the natural log of mean dietary adequacy of protein, Ca, and vitamin B12 for children 12-48 months (at baseline) in consumer households?

The study population will include dairy vendors operating in the informal sector (businesses selling unpackaged or not-formally processed milk to individual consumers; this includes raw, boiled and unpacked pasteurized milk) in the study areas and consumer households that purchase most of their weekly milk from those vendors. The unit of randomization is a cluster of 1 to 5 vendors and the households consuming milk from those vendors. Clusters are identified using a hybrid approach based on a computer-based algorithm informed by the GPS locations of the informal milk vendors in the target areas. The resulting clusters ensure that vendors in one cluster are located at least 250m away from any vendor in a different cluster. Study clusters will be randomly assigned to one of two arms:

1. Treatment arm: Training, certification, and marketing scheme for milk vendors.
2. Control arm: Delayed intervention (implemented after endline survey). Study vendors in the intervention (treatment) clusters will be offered the possibility to participate in a 12-15hr training. Trainings will be offered free of charge. Upon completion of the endline survey, vendors in the control clusters will also be offered the training, which will follow the same format as the one used in the intervention clusters. The training will be offered a few hours per day over 5-days to accommodate vendors' time constraints, which we expect to be more severe for female vendors. The trainings will be given by business development service (BDS) providers. BDS correspond to a "wide range of non-financial services provided by public and private suppliers (BDS providers) to entrepreneurs to help them operate efficiently and to grow their business with the broader purpose of contributing to economic growth, employment generation and poverty alleviation" (Kimando, 2012). The Kenyan register of BDS providers will be used to identify available BDS providers. The selected BDS will receive a full training course, covering the intervention content and specific teaching methods to be used during the training of vendors.

The study will include 142 vendor clusters (with a minimum number of vendors per cluster of one and a maximum of five), 240 vendors and 852 households at baseline. For the health outcome, the study will be powered to detect a 0.4 standard deviation difference between the natural log of TBC in the treatment and control groups. This equates roughly to a 20 percentage point increase in the proportion of vendors selling milk meeting EAS one year after the intervention, off of a proportion of 37% in the data we collected in the study areas in 2017. For the nutrition outcomes, the study will be powered to detect a change in the natural log of mean dietary adequacy of Ca, protein, and vitamin B12 that corresponds to a daily increase of 75gr of milk (0.5 cups) consumed per child. This is one-third of the median daily milk consumption for children 24-48 months of age in the MilkMarkets data collected in Dagoretti in 2017.

Randomization of vendor cluster to treatment or control arm will be conducted immediately after completion of the baseline surveys for vendors and consumer households, and hence post-consent. After randomization, vendors in clusters allocated to the intervention will be contacted, informed of the training schedules available in their ward, and offered the possibility to attend 1 of up to 3 scheduled training options. Vendors in the control clusters will be informed that they will be given the option to participate in the trainings one year later.

Selection and recruitment of vendors - From the full list of identified clusters, we will randomly select the 142 to meet the study sample size requirements. In each cluster, a minimum of 1 and a maximum of 5 vendors will be recruited.

Selection and recruitment of households - For each participating cluster, we will recruit up to 6 consumer households that meet our inclusion criteria. Each recruited vendor will be given a small add to display in their business/premise advertising the study and inviting interested consumers to register interest to participate in the study by providing their name and telephone number in a registration form. Vendors will be encouraged to bring the study to the attention of their customers. The information will be kept at the vendor's premise for up to 10 days and then collected by field workers. Registered consumers will be contacted and information collected to check their eligibility (see criteria above). If not enough eligible households were identified, a second approach to recruitment will be used. A field worker will spend 2-3 hours in the morning or the evening of a given day at the recruited vendor's premise and approach customers that purchase liquid unprocessed milk during this time period. A brief set of questions will be asked to confirm whether the consumer household meets our inclusion criteria. If it does, the study will be presented and interest to participate in the study will be recorded. Basic contact details will be obtained to facilitate follow up. After identification of all eligible households in the cluster, 6 households will be randomly selected to participate in the study aiming at achieving equal number of household per vendor(whenever there is more than 1 vendor in a cluster) and ensuring there is at least one household per vendor in each cluster.

Selection of the index child - In each recruited household one child 12 months to 48 months of age will be selected. If only one child falls into this age window at the time of baseline, this child will be the index child. In case there are multiple children in the household meeting the age criterion, the index child will be randomly selected manually or by the computer-assisted personal interview software.

A baseline survey and an endline survey will be conducted in recruited vendors and households prior to the intervention (baseline) and 12 months after baseline (endline). The questionnaire to vendors will gather information on the following three elements: (i) milk hygiene and handling practices of daily operations, including sourcing of milk, equipment available and use of quality testing; (ii) business performance, recording milk volumes purchased/sold, expenditures, revenues and cost of equipment; (iii) women's empowerment in their business and related household gender dynamics. In addition, two un-announced visits to the participating vendors will be conducted between the intervention and the enline survey, where observable features on milk hygiene and handling will be recorded through a short questionnaire. These two mid-term visits will allow for collection of information on business performance indicators and any unexpected negative consequences from participation in the study. In households, questionnaires will record the following information (i) household food expenditure, with focus on milk products; (b) milk consumption, handling and hygiene practices; (c) a 24hr dietary recall for the selected child 12-48 months at baseline; (d) presence of diarrhea in the past 7 days (diarrhea understood as one or more days having at least 3 loose stools/day).

At baseline, endline, and at the 2 unannounced visits, up to 100ml of milk sold by participating vendors will be bought. Samples will be tested for total bacterial counts (TBC), enumeration of enterobacteriaceae and presence and enumeration of coagulase positive staphylococci. For vendors in the intervention clusters, results of the laboratory analysis and feedback on milk hygiene practices will be communicated after each testing.

The "multiple-pass" 24hr recall method will be used. This approach uses a special method to help the primary caretaker, usually the mother, of a child remember what was consumed and ensure that enumerators do not miss important information. Using the 24hr form, enumerators review the day's food and drink several times with the primary caretaker of the child. Each time, or "pass" more detailed information is added to the recall form, thus reducing the probability that foods are omitted. A detailed 24hr recall protocol has been developed. Length/height and weight of the selected child and his/her mother will be recorded.

The process evaluation will examine the primary inputs, processes, outputs, and outcomes along the program impact pathway to determine the "how" and "why" of program impact. The scope of the process evaluation is limited to providing a qualitative assessment of issues related to program implementation and delivery. A combination of random and purposive sampling techniques will be used for the process evaluation. Quantitative data will be collected through precoded questionnaires. Qualitative data will be collected through semi-structured continuous observations of program activities, semi-structured individual qualitative interviews with implementation staff and beneficiaries, and group free listing with beneficiaries.

A scientific advisory committee has been set up, formed of 3 individuals external to the research team and to the project partner institutions. The Committee will revise and provide feedback on the study protocol and the study research tools (questionnaires, consent forms, …), as well as conduct data monitoring for selected indicators. The Committee will select a chair for the duration of the study, who will convene meetings as required based on the outcomes of the monitoring.

ELIGIBILITY:
Inclusion Criteria (dairy vendors):

* Operate in the informal dairy sector (i.e. selling unpacked milk, not-formally processed milk) at least 5 days per week and indicates (at baseline) an intention to remain in the business at least for the next 12 months.
* Operate a milkbar (i.e. business exclusively selling dairy products and eggs), a shop/kiosk (i.e. licensed for selling other products) or be a street vendor (i.e. not selling in a fixed building structure but in a specific location along the street).
* Sell milk directly to individual consumers/households.

Inclusion Criteria (households):

* Buying unpacked milk
* Meet at least 50% of its weekly milk needs with unpacked milk from a recruited vendor.
* Have at least one child 12 to 48 months of age at the time of recruitment.

Inclusion Criteria (children):

* 12 to 48 months of age at baseline

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Health outcome: total bacterial count (TBC) per mL of milk sold by vendors | 12 months after baseline
  Total bacterial count represents the number of viable aerobic bacteria present in one mL of milk and reflects the hygienic handling of milk from production to the point of testing. It is a well-established food hygiene indicator and the primary milk safety indicator in the East African Standards for Raw Milk. While it is a good indicator of the sanitary quality of the milk, it does not directly correlate to the presence of pathogens or toxins in a food product. However, food products with high TBC can be reasonably assumed to carry health hazards. Given that the distributions of TBC in food products are highly skew, we will analyze this outcome with an appropriate log transformation, which is likely to be the natural log (which is the most commonly used log transformation when analyzing TBC and the one considered for power calculations in this study) or a stronger fractional power of root.
Nutrition outcome: mean dietary adequacy of protein, Ca, and vitamin B12 in children 12-48 months at baseline | 12 months after baseline
  Milk contains protein and calcium and is a good source of vitamin B12. The promotion of milk by vendors in the treatment arm is expected to increase milk consumption in children, but it may also lead to reduced intake of other nutrient-dense foods. We will assess the dietary adequacy of these three nutrients in the overall diet. The outcome will be constructed by first calculating the dietary adequacy for each key nutrient (i.e. protein, calcium, and vitamin B12). Nutrient adequacy is defined as the observed nutrient intake divided by the age-specific nutrient requirement. We will then calculate the mean adequacy across all three nutrients for each individual. We expect the distribution of mean dietary adequacy to be positively skew and we will therefore use the natural log of mean dietary adequacy in the analysis or a stronger fractional power of root, if required

SECONDARY OUTCOMES:
Differential treatment effect on total bacterial count in milk | 4, 8 and 12 months after baseline
  The difference in the magnitude of treatment effect on total bacterial count over 1 year of monitoring, tested at 3 time points.
Enterobacteriaceae count in milk | 12 months after baseline
  Number of enterobacteriaceae per mL of milk. Enterobacteriaceae group includes coliforms, Salmonella, Shigella and Yersinia, among others
Coagulase positive staphylococci (CPS) in milk | 12 months after baseline
  Proportion of vendors having milk with <1 coagulase positive staphylococci (CPS) per mL
Business profitability | 12 months after baseline
  increase in milk-related monthly profits (revenues minus costs)
Mean women's empowerment index-score of vendors and their spouses | 12 months after baseline
  The overall mean women's empowerment index-score (WEAI) in vendors and their spouses and the mean score in 2 specific domains of empowerment
Child linear growth | 12 months after baseline
  Height-for-age difference and prevalence of stunting (defined as having a height-for-age Z-score below -2SD)
Child weight | 12 months after baseline
  Child weight and prevalence of wasting (defined as having a weight-for-height Z-score below -2 SD)
Child milk intake | 12 months after baseline
  Grams of milk consumed per day
Child dietary adequacy | 12 months after baseline
  mean probability of adequacy (MPA) in micronutrient intake and probability of adequacy of iron, zinc and vitamin A
Child acute diarrhea | 12 months after baseline
  Presence of diarrhea in the past 7 days (with diarrhea defined as one or more consecutive days with at least 3 loose stools/day)

OTHER OUTCOMES:
Dairy vendors milk handling and business practices | 12 months after baseline
  Proportion of households improving milk handling and business practices
Household's milk handling knowledge and practices | 12 months after baseline
  Proportion of households improving milk handling knowledge and practices
Mean dimension-specific women's empowerment index-score of vendors and their spouses | 12 months after baseline
  Mean women's empowerment index-score in additional domains of empowerment

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Alonso, PhD, Principal Investigator — The International Livestock Research Institute (ILRI)
Locations (1):
- International Livestock Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No
IDP will be treated in high confidentiality given the sensitivity of the information. Some of the participants in the study may be operating in an ambiguous legal situation and their confidentiality must be preserved both during and after the study.